CLINICAL TRIAL: NCT04973410
Title: FLOW 3 - The Association Between Catheter-based Coronary Flow and Resistance and 15O-H2O Positron Emission Tomography Scan-based Absolute Myocardial Blood Flow in the Coronary Artery Territory.
Brief Title: The Association Between Catheter-based Coronary Flow and Resistance and 15O-H2O Positron Emission Tomography Scan
Acronym: FLOW3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, Clinical Associate Professor, Aarhus University Hospital Skejby
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-239-19
Record Dates: First submitted 2021-03-17; First posted 2021-07-22 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: Thermodilution method; FFR; IMR; CFR; PET; Myocardial Blood Flow
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): FFR negative/non-significant (>0.80) and IMR negative (<25)
  Interventions: Diagnostic Test: Coronary Physiology; Diagnostic Test: 15O-H2O-PET scan
- Group B (Other): FFR negative/non-significant (>0.80) and IMR positive (>25)
  Interventions: Diagnostic Test: Coronary Physiology; Diagnostic Test: 15O-H2O-PET scan

INTERVENTIONS:
Diagnostic Test: Coronary Physiology — Invasive coronary physiology measurements during diagnostic CAG with thermodilution method with the CoroFlow® (Coroventis, Uppsala, Sweden)
  Other Names: IMR, FFR, CFR
Diagnostic Test: 15O-H2O-PET scan — Myocardial blood flow (MBF) measured with oxygen-15 (O-15) labelled water used as a tracer molecule with positron emission tomography (PET)

SUMMARY:
Aims

1. To assess the correlation between absolute flow and resistance assessed by catheter-based thermodilution technique using CoroFlow®-system and myocardial blood flow (MBF) measured by positron emission tomography (PET) and the tracer [15O] labeled water ([15O]H2O) (15O-H2O PET)
2. To assess the correlation between impaired MBF measured with 15O-H2O PET and negative fractional flow reserve (FFR) and index of microvascular resistance (IMR) level.

Hypothesis:

In patients with angina pectoris and reduced MBF measured with 15O-H2O PET but no hemodynamic significant stenosis (FFR > 0.80), the IMR is >25 measured with continuous thermodilution indicating microcirculatory dysfunction.

Methods:

We include patients with angina pectoris and suspected coronary disease based on a cardiac-computerised tomography (CT) scan. Patients are then referred to an 15O-H2O PET (rest and stress) and then a diagnostic invasive coronary angiography (ICA) with physiological assessment.

DETAILED DESCRIPTION:
Background Computer tomography coronary angiography (CTCA) is a purely an anatomical scan and can be insufficient in assessing the significance of a coronary stenosis. The latest European guidelines recommend that, as a supplementary study after heart CT and before invasive coronary angiography (ICA), a myocardial perfusion study is performed to avoid unnecessary invasive procedures.

Several PET flow tracers are available, but 15O-H2O is considered the gold standard for quantification of regional myocardial perfusion since 15O-H2O is a freely diffusible tracer. 15O-water PET has been validated for measure perfusion in myocardium.

15O-H2O is an inert radiopharmaceutical of oxygen-15 (O-15) labelled water used as a tracer molecule with positron emission tomography (PET). Upon administration, 15O-H2O is freely diffusible and its distribution, as well as its clearance, are completely dependent on the rate of blood flow. 15O-H2O PET imaging is golden standard for measure tissue perfusion including myocardial perfusion. The PET agent 15O-H2O has a very short half-life of about 2 minutes thereby allowing for multiple, serial measurements. Two recent studies have described the diagnostic accuracy of 15O-H2O PET in comparison to coronary angiography.

In both studies, 15O-H2O PET had a sensitivity of 87-95%; specificity was at least 84%. The study by Danad et al7 is the largest published series to date. A recently published single-center study compared 15O-H2O PET to imaging using 99mTc and found superior performance characteristics for the 15O-H2O PET, relative to a truth standard of ICA with fractional flow reserve (FFR).

Fractional flow reserve (FFR) is defined as the maximum achievable blood flow that can still be maintained to myocardium despite the stenosis. Also described as the ratio between the pressure distal to the stenosis (Pd) and the pressure proximal (Pa) to the lesion during hyperemia.

In randomized trials the benefits of FFR measurements was established by comparing FFR-guided PCI plus medical therapy with just medical therapy. This showed that patients with stable coronary artery disease will benefit from FFR-guided PCI plus medical therapy in that the risk of needing urgent revascularization will be smaller.9 Randomized trials also show that if an intermediate coronary stenosis - not functionally significant - is measured to have an FFR ≥0.75, the risk of infarction from that stenosis is less than 1 %. Therefore, these patients will not benefit from PCI.10 This makes FFR an important tool for assessing which patients could benefit from a PCI and which are better off with the best medical therapy available. However, it only describes the flow of the epicardial arteries. FFR value may be non-significant (>0.80) while the patient may still have angina. This may be due to microvascular disease. The evaluation of the microvascular status when the FFR indicates non-obstructive disease (>0.80) currently has IIa indication in the ECS guidelines.

Thermodilution method with the CoroFlow® (Coroventis, Uppsala, Sweden) from which coronary flow reserve and microvascular resistance can be calculated alongside the FFR value. This gives us opportunity to study coronary microcirculatory dysfunction and is believed to be common in patients with angina and no significant disease in the epicardial arteries. However, there is a gap in evidence in terms of finding the best method to conduct quantitative assessment of the microcirculatory system independently of epicardial stenoses.13 Furthermore, the combination of coronary flow reserve and microvascular resistance measured by invasive thermodilution method (CoroFlow®-system) has not previously been compared to myocardial blood flow (MBF) measured with the golden standard 15O-H2O PET.

Methods:

Physiological assessment protocol The ICA is performed according to present clinical guidelines through femoral or radial ar-tery. Prior to the coronary angiography, the operator administrates 250 μg of intra-coronary nitroglycerine. Anticoagulation (5,000 IU heparin) is administrated before the measure-ment.

Coronary physiological assessment is performed in all vessels (left anterior descending (LAD), right coronary artery (RCA) and the circumflex artery (CX)) with the thermodilution method measuring fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microcirculatory resistance (IMR).

The guidewire equipped with a pressure and temperature sensor (PressureWire X, Abbott, IL) is passed through the guiding catheter. The operator infuses saline at room temperature 3 times in rest. Hyperaemia is then induced with adenosine was infused intravenously (140 mg/kg/min, then the operator infuses saline at room temperature at hyperaemia.

The Coroventis system is used as pressure measuring software. Routine checks are made to ensure that 'drift' does not occur after the recordings. Drift value of ≤ ±0.02 is accepted.

Protocol 15O-H20 PET Study participants will be instructed to avoid all caffeine-containing drinks and foods such as coffee, chocolate, cola, banana and tea for at least 24 hours prior to the planned admin-istration of adenosine.

Quantitative myocardial perfusion at rest and during hyperemia will be measured using 2 injections (rest & stress) of 400 MBq of 15O-H2O.

After an initial scout CT scan to localize the heart, a low-dose CT for attenuation correction (CTAC) of the subsequent PET emission data is performed. Following the CTAC, the rest and stress PET scans will be performed in that order.

Rest scan: A PET list mode acquisition of 4 minutes in duration should be started just before the intravenous injection of 400 MBq of 15O-H2O from a water generator (MedTrace P3 system). List mode data is reconstructed with ECG-signal to an 8-bin ECG-gated blood pool image of the first pass (0-50 seconds after injection) and a dynamic data set of 22 frames from 0-4 minutes after injection.

Stress scan: Pharmacological stress is induced by infusion of adenosine intravenously at a standard rate of 140µg/kg/min. Following 2 minutes of adenosine injection, vasodilation is known to reach a steady state, a second dose of 15O-H2O (400 MBq) is injected, and a new PET scan is performed like the rest scan (list mode imaging initiated before the bolus IV injection).

During both acquisitions and the stress test, heart rate and blood pressure as well as any ECG related abnormalities is monitored.

Data from rest and stress 15O-H2O PET scans will be analyzed using the aQuant software.

Statistics and power calculations:

Student's t-test will be used for continuous variables and non-parametric test for categorical variables. The diagnostic performance of 15O-H2O PET is assessed by Bland-Altmann plot and receiver operative curves. The result quality will be assessed according to the P-value (P>0.05) significance between low and high IMR groups. With a standard deviation of 10, mean difference of 15, power of 80 % and alpha value of 0.05, n=22 patients in total are needed. To accommodate for drop outs 40 patients i.e. 20 in two groups are included. In group A will be patients with a non-significant FFR value (<0.80) and an IMR value indicating no microcirculatory dysfunction (IMR <25). In group B will be patients with a non-significant FFR value (<0.80) and an IMR value indicating microcirculatory dysfunction (IMR ≥25).

Publication of results Results, positive, neutral as well as negative or inconclusive, will be published in an international cardiovascular journal without delay. Publication and author issues are decided by the steering committee on basis of general involvement in the study (drafting of protocol, core lab. function, end point committee membership, etc.) and of number of included patients. The funding companies have no influence on study design, study conduct, analysis, interpretation and reporting of derived results.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to diagnostic ICA after heart-CT
* Able to provide an informed consent.
* Age ≥ 18 years

Exclusion Criteria:

* PCI, CABG, POBA or already acknowledge ischemic heart disease
* Acute coronary disease or AMI
* COPD or Asthma
* Pregnancy and breast breeding
* Contraindications to adenosine (severe asthma, complicated AV block, critical aortic stenosis, severe cardiac arrhythmias, severe valve diseases).
* Renal impairment with estimated glomerular filtration rate (eGFR) <40 ml / min.
* Allergy to X-ray contrast agents or severe metabolic disease.
* Donor heart, mechanical heart, or mechanical heart pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity for absolute myocardial blood flow measured by 15O-H2O PET in detection of coronary microcirculatory diseases measured by index of microcirculatory index (IMR) | From the 15O-H2O PET scan to the coronary physiology assessment during ICA, up to 1 week.
  Sensitivity, specificity for absolute myocardial blood flow measured by 15O-H2O PET in detection of coronary microcirculatory diseases measured by index of microcirculatory index (IMR) during catheter-based thermodilution technique.
  The diagnostic performance of 15O-H2O PET between low and high IMR groups
The diagnostic performance of 15O-H2O PET between low and high IMR groups | From the 15O-H2O PET scan to the coronary physiology assessment during ICA, up to 1 week.
  positive predictive value (PPV), negative predictive value (NPV) for absolute myocardial blood flow measured by 15O-H2O PET in detection of coronary microcirculatory diseases measured by index of microcirculatory index (IMR) during catheter-based thermodilution technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pakkal M, Raj V, McCann GP. Non-invasive imaging in coronary artery disease including anatomical and functional evaluation of ischaemia and viability assessment. Br J Radiol. 2011 Dec;84 Spec No 3(Spec Iss 3):S280-95. doi: 10.1259/bjr/50903757. PMID 22723535
- [Background] Wood DJ, Mason JB, Chapman HM. Scrapie scruples. N Z Vet J. 1978 Jul;26(7):190-1. doi: 10.1080/00480169.1978.34537. No abstract available. PMID 278924
- [Background] Huang SC, Schwaiger M, Carson RE, Carson J, Hansen H, Selin C, Hoffman EJ, MacDonald N, Schelbert HR, Phelps ME. Quantitative measurement of myocardial blood flow with oxygen-15 water and positron computed tomography: an assessment of potential and problems. J Nucl Med. 1985 Jun;26(6):616-25. PMID 3873525
- [Background] Bergmann SR, Fox KA, Rand AL, McElvany KD, Welch MJ, Markham J, Sobel BE. Quantification of regional myocardial blood flow in vivo with H215O. Circulation. 1984 Oct;70(4):724-33. doi: 10.1161/01.cir.70.4.724. PMID 6332687
- [Background] Berti V, Sciagra R, Neglia D, Pietila M, Scholte AJ, Nekolla S, Rouzet F, Pupi A, Knuuti J. Segmental quantitative myocardial perfusion with PET for the detection of significant coronary artery disease in patients with stable angina. Eur J Nucl Med Mol Imaging. 2016 Jul;43(8):1522-9. doi: 10.1007/s00259-016-3362-0. Epub 2016 Mar 18. PMID 26993310
- [Background] Kajander S, Joutsiniemi E, Saraste M, Pietila M, Ukkonen H, Saraste A, Sipila HT, Teras M, Maki M, Airaksinen J, Hartiala J, Knuuti J. Cardiac positron emission tomography/computed tomography imaging accurately detects anatomically and functionally significant coronary artery disease. Circulation. 2010 Aug 10;122(6):603-13. doi: 10.1161/CIRCULATIONAHA.109.915009. Epub 2010 Jul 26. PMID 20660808
- [Background] Danad I, Uusitalo V, Kero T, Saraste A, Raijmakers PG, Lammertsma AA, Heymans MW, Kajander SA, Pietila M, James S, Sorensen J, Knaapen P, Knuuti J. Quantitative assessment of myocardial perfusion in the detection of significant coronary artery disease: cutoff values and diagnostic accuracy of quantitative [(15)O]H2O PET imaging. J Am Coll Cardiol. 2014 Oct 7;64(14):1464-75. doi: 10.1016/j.jacc.2014.05.069. PMID 25277618
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Background] Corcoran D, Young R, Adlam D, McConnachie A, Mangion K, Ripley D, Cairns D, Brown J, Bucciarelli-Ducci C, Baumbach A, Kharbanda R, Oldroyd KG, McCann GP, Greenwood JP, Berry C. Coronary microvascular dysfunction in patients with stable coronary artery disease: The CE-MARC 2 coronary physiology sub-study. Int J Cardiol. 2018 Sep 1;266:7-14. doi: 10.1016/j.ijcard.2018.04.061. Epub 2018 Apr 19. PMID 29716756
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Xaplanteris P, Fournier S, Keulards DCJ, Adjedj J, Ciccarelli G, Milkas A, Pellicano M, Van't Veer M, Barbato E, Pijls NHJ, De Bruyne B. Catheter-Based Measurements of Absolute Coronary Blood Flow and Microvascular Resistance: Feasibility, Safety, and Reproducibility in Humans. Circ Cardiovasc Interv. 2018 Mar;11(3):e006194. doi: 10.1161/CIRCINTERVENTIONS.117.006194. PMID 29870386
- [Background] Luo C, Long M, Hu X, Huang Z, Hu C, Gao X, Du Z. Thermodilution-derived coronary microvascular resistance and flow reserve in patients with cardiac syndrome X. Circ Cardiovasc Interv. 2014 Feb;7(1):43-8. doi: 10.1161/CIRCINTERVENTIONS.113.000953. Epub 2014 Jan 7. PMID 24399243
- See also: Fractional Flow Reserve (FFR) - Shown To Improve Patient Outcomes And Reduce Costs. October 2013 — https://www.radcliffecardiology.com/articles/fractional-flow-reserve-ffr-shown-improve-patient-outcomes-and-reduce-costs